CLINICAL TRIAL: NCT05161689
Title: Addressing the Continuum of Care Among High-risk Thai Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: University of California, San Francisco (Other); University of Malaya (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH119015 (NIH); R01MH119015 (NIH)
Record Dates: First submitted 2021-11-03; First posted 2021-12-17 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: HIV/AIDS; STD
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: The community-based, multilevel and theory-based intervention diffuses social support and empowers the YMSM community in order to establish social norms supportive of risk reduction and biannual HIV testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mpowerment-based intervention (Experimental): YMSM in this arm may be exposed to a multicomponent, multi-level, community mobilization, combination intervention to address the entire HIV Continuum of Prevention and Care.
  Interventions: Behavioral: HUG-M+
- Standard of care (No Intervention): YMSM in this arm will not be exposed to the intervention.

INTERVENTIONS:
Behavioral: HUG-M+ — A multicomponent, multi-level, community mobilization, combination intervention (HUG-M+) to address the entire HIV Continuum of Prevention and Care.
  Arms: Mpowerment-based intervention

SUMMARY:
Young Thai men who have sex with men (YMSM) are at high risk for HIV. However, the Thailand National HIV Strategy does not adequately cover HIV prevention for YMSM using specific methods relevant to them, and instead uses a one-size-fits all approach. Partnering with the Thailand Ministry of Public Health (MOPH), the proposed study seeks to finalize, implement and evaluate a multicomponent, multi-level, community mobilization, combination intervention (HUG-M+) to address the entire Continuum of Prevention and Care. The investigators propose to test the efficacy of this approach by conducting research in two Northeastern Thai cities, one randomized to the intervention condition, which will receive HUG-M+ and the other to the control condition, where standard of care will be provided. If HUG-M+ is found to be efficacious, it might be scaled up, with the support of the MOPH, to other regions in Thailand, elsewhere in Asia and the US.

DETAILED DESCRIPTION:
The HIV epidemic in Thailand is escalating among young men who have sex with men (YMSM). Particularly, HIV prevalence among YMSM is estimated to be 10-15% in Northeastern Thailand. Obviously high risk sexual behavior is occurring, and the uptake of HIV testing remains low even though free testing services are offered by public clinics. Despite provision of free antiretroviral treatment (ART) by the government, less than 25% of HIV-positive YMSM (HIV+YMSM) are retained in care, suggesting very few have achieved viral suppression. The suboptimal access to HIV testing and treatment services among YMSM pose tremendous challenge in much needed prevention efforts to improve linkage to care and achieve individual and community viral suppression to prevent onward HIV transmission. Community mobilization and an empowerment approach that targets barriers at individual, social/community, and health systems levels are needed to improve access to prevention and treatment services, including sexual risk reduction, HIV testing, and linkage and engagement in the care continuum (CC). Based on a cultural adaptation of the evidence-based Mpowerment intervention, we developed and piloted HUG-M, a multilevel, theory-based intervention that diffuses social support and empowers the YMSM community in order to establish social norms supportive of risk reduction and biannual HIV testing. HUG-M was acceptable to YMSM in a prior pilot study, feasible to implement, and has the potential to increase HIV testing and decrease sexual risk behavior. The proposed study will test a community mobilization, multi-level intervention in two well-matched cities in Northeastern Thailand. The project's aims are: (1) to finalize and manualize HUG-M+, a community mobilization, multicomponent, multi-level, combination intervention that focuses on the entire Continuum of Prevention and Care, (2) to implement HUG-M+ for 2 years in collaboration with the Thailand Ministry of Public Health (MOPH) clinics that provide HIV testing and treatment, and (3) to evaluate the pilot efficacy of HUG-M+ in decreasing sexual risk behavior; increasing HIV testing to at least biannually; and increasing prompt, sustained engagement in care among men living with HIV by (a) longitudinal cohorts of YMSM in two cities in Northeastern Thailand; oversampling HIV+YMSM, which will provide data on the CC including sexual risk behavior; anal bacterial STIs; HIV testing frequency; and engagement in care among HIV+YMSM; and (b) longitudinal public health data, already collected by the MOPH, which include CD4 and viral load data for HIV patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 15-29 years at cohort baseline
* Self-reported male gender
* Self-reported having had anal sex with another man in the past 12 months
* Speak, read and write Thai
* Thai citizenship
* Resident of the assessment city for the next 2 years (live, work or go to school)

Exclusion Criteria:

* Do not consent to urine testing or anal swab
* Not willing to give contact information for follow-up assessments

Ages: 15 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Since this study is focusing on an HIV key population, namely men who have sex men, participants need to be biological males and identify as males.
Enrollment: 636 (Actual)
Dates: Start 2021-11-27 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Guadamuz, PhD, Principal Investigator — Mahidol University
Locations (2):
- Thailand (2):
  - M-Health Office Maha Sarakham, Maha Sarakham
  - M-Health Office Ubon, Ubon Ratchathani

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Samoh N, Peerawaranun P, Jonas KJ, Lim SH, Wickersham JA, Guadamuz TE. Willingness to Use HIV Self-Testing With Online Supervision Among App-Using Young Men Who Have Sex With Men in Bangkok. Sex Transm Dis. 2021 Mar 1;48(3):e41-e44. doi: 10.1097/OLQ.0000000000001271. PMID 32842048
- [Background] Guadamuz TE, Goldsamt LA, Boonmongkon P. Consent Challenges for Participation of Young Men Who Have Sex With Men (YMSM) in HIV Prevention Research in Thailand. Ethics Behav. 2015 Mar;25(2):180-195. doi: 10.1080/10508422.2014.949721. PMID 25750498
- [Background] Guadamuz TE, Boonmongkon P. Ice parties among young men who have sex with men in Thailand: Pleasures, secrecy and risks. Int J Drug Policy. 2018 May;55:249-255. doi: 10.1016/j.drugpo.2018.04.005. Epub 2018 Apr 23. PMID 29691128
- [Background] Guadamuz TE, McCarthy K, Wimonsate W, Thienkrua W, Varangrat A, Chaikummao S, Sangiamkittikul A, Stall RD, van Griensven F. Psychosocial health conditions and HIV prevalence and incidence in a cohort of men who have sex with men in Bangkok, Thailand: evidence of a syndemic effect. AIDS Behav. 2014 Nov;18(11):2089-96. doi: 10.1007/s10461-014-0826-8. PMID 24989128
- [Background] Kongjareon Y, Samoh N, Lim SH, Peerawaranun P, Jonas KJ, Guadamuz TE. Group sex, suicidality and online partners: implications for HIV and suicide prevention: a short report. AIDS Care. 2020 Aug;32(8):954-958. doi: 10.1080/09540121.2020.1734174. Epub 2020 Mar 12. PMID 32160793

RESULTS

PARTICIPANT FLOW:
Groups:
- Mpowerment-based Intervention: Young men who have sex with men (YMSM) in this arm may be exposed to a multicomponent, multi-level, community mobilization, combination intervention to address the entire HIV Continuum of Prevention and Care.
  HUG-M+: A multicomponent, multi-level, community mobilization, combination intervention (HUG-M+) to address the entire HIV Continuum of Prevention and Care.
Period: Overall Study
Arm/Group | Mpowerment-based Intervention | Standard of Care
Started | 318 | 318
Completed 6 Months Follow-up | 259 | 236
Completed 12 Months Follow-up | 234 | 231
Completed 18 Months Follow-up | 218 | 223
Completed 24 Months Follow-up | 187 | 205
Completed | 187 | 205
Not Completed | 131 | 113

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mpowerment-based Intervention | Standard of Care | Total
Number analyzed (Participants) | 318 | 318 | 636
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 56 | 80 | 136
  Between 18 and 65 years | 262 | 238 | 500
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.1 (3.1) | 20.1 (2.6) | 20.6 (2.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Self-Identified Sexual/Gender Identity: Transwomen who are Biologically Male | 3 | 11 | 14
  Self-Identified Sexual/Gender Identity: Males who have sex with Men | 285 | 292 | 577
  Self-Identified Sexual/Gender Identity: Bisexual Males | 30 | 15 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Thai | 318 | 318 | 636
Region of Enrollment [Number; unit: participants]
  Thailand | 318 | 318 | 636
Self-Reported Last HIV Testing Date [Count of Participants; unit: Participants]
  Never tested | 141 | 178 | 319
  More than 12 months ago | 52 | 63 | 115
  7-12 months ago | 33 | 29 | 62
  ≤ 6 months ago | 92 | 48 | 140
HIV status data from Ministry of Public Health national database [Count of Participants; unit: Participants]
  HIV-positive | 76 | 26 | 102
  HIV-negative | 126 | 169 | 295
  Not Found in System | 116 | 123 | 239
Condom use consistency during anal sex with men over the past 6 months [Count of Participants; unit: Participants]
  Never | 3 | 9 | 12
  Less than half the time | 9 | 7 | 16
  About half the time | 14 | 8 | 22
  More than half the time | 30 | 39 | 69
  Every time | 76 | 59 | 135
  Did not have anal sex with men in the past 6 months | 186 | 196 | 382
STI Prevalence (Chlamydia and Gonorrhea) [Count of Participants; unit: Participants] | 58 | 53 | 111
Participation in group sex activities (ever) [Count of Participants; unit: Participants] | 46 | 61 | 107
Participant has given or received items or opportunities in exchange for sex [Count of Participants; unit: Participants]
  Yes, I was the one receiving money, things, or opportunities | 36 | 41 | 77
  Yes, I was the one giving money, things, or opportunities | 7 | 2 | 9
  Yes, I have both given and received money, things, or opportunities | 10 | 6 | 16
  No | 265 | 269 | 534
Participant has agreed to meet someone contacted online (via app or website) for sex [Count of Participants; unit: Participants] | 183 | 191 | 374
Participant has had anal sex with a man while under the influence of drugs or alcohol [Count of Participants; unit: Participants] | 77 | 94 | 171
Number of Participants with Depression (CES-D-10) [Count of Participants; unit: Participants] — Depression was assessed using the 10-item Center for Epidemiologic Studies Depression Scale (CES-D-10), a validated screening tool for depressive symptoms. Each item is rated on a 4-point Likert scale ranging from 0 ("Rarely or none of the time") to 3 ("All of the time"). The total score ranges from 0 to 30, with higher scores indicating more severe depressive symptoms. A total score of ≥10 was used as the cut-off to classify participants as having depression. The reported outcome reflects the number and percentage of participants meeting this cut-off.
  Participants | 110 | 114 | 224
Number of Participants at Risk of Suicide (SBQ-R) [Count of Participants; unit: Participants] — Suicidal risk was assessed using the Suicide Behaviors Questionnaire-Revised (SBQ-R), a validated screening tool for suicidal thoughts and behaviors. The SBQ-R includes 4 items assessing (1) lifetime suicidal ideation and/or attempts, (2) frequency of suicidal ideation in the past 12 months, (3) threats of suicide attempts, and (4) self-reported likelihood of future suicidal behavior. Total scores range from 3 to 18, with higher scores indicating greater risk. Participants with a total score of ≥7 were classified as being at risk of suicide. The reported outcome reflects the number and percent
  Participants | 65 | 79 | 144

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of HIV Testing in the Past 6 Months Among YMSM at Baseline
Description: Number of Participants who answered "yes" to the question if they have tested in the past 6 months
Time Frame: Assessed at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Mpowerment-based Intervention | Standard of Care
Number analyzed (Participants) | 318 | 318
Participants | 92 | 48

2. Primary Outcome: Prevalence of HIV Testing in the Past 6 Months Among YMSM at 6 Months
Description: Number of Participants who answered "yes" to the question if they have tested in the past 6 months
Time Frame: Assessed at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mpowerment-based Intervention | Standard of Care
Number analyzed (Participants) | 259 | 236
Participants | 114 | 80

3. Primary Outcome: Prevalence of HIV Testing in the Past 6 Months Among YMSM at 12 Months
Description: Number of Participants who answered "yes" to the question if they have tested in the past 6 months
Time Frame: Assessed at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mpowerment-based Intervention | Standard of Care
Number analyzed (Participants) | 234 | 231
Participants | 104 | 98

4. Primary Outcome: Prevalence of HIV Testing in the Past 6 Months Among YMSM at 18 Months
Description: Number of Participants who answered "yes" to the question if they have tested in the past 6 months
Time Frame: Assessed at 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mpowerment-based Intervention | Standard of Care
Number analyzed (Participants) | 218 | 223
Participants | 96 | 96

5. Primary Outcome: Prevalence of HIV Testing in the Past 6 Months Among YMSM at 24 Months
Description: Number of Participants who answered "yes" to the question if they have tested in the past 6 months
Time Frame: Assessed at 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mpowerment-based Intervention | Standard of Care
Number analyzed (Participants) | 187 | 205
Participants | 61 | 77

6. Primary Outcome: Prevalence of Condomless Anal Sex in the Past 6 Months Among YMSM at Baseline
Description: Participants will answer a yes/no question if they engage in condomless anal intercourse (CAI) with non-primary or primary partners who are serodiscordant or of unknown serostatus, nonmonogamous, or who have been primary partners less than 6 months.
Time Frame: Assessed at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Mpowerment-based Intervention | Standard of Care
Number analyzed (Participants) | 318 | 318
Participants | 56 [10.5 to 17.0] | 63 [16.9 to 19.3]

7. Primary Outcome: Prevalence of Condomless Anal Sex in the Past 6 Months Among YMSM at 6 Months
Description: as for outcome 6
Time Frame: Assessed at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mpowerment-based Intervention | Standard of Care
Number analyzed (Participants) | 259 | 236
Participants | 37 | 42

8. Primary Outcome: Prevalence of Condomless Anal Sex in the Past 6 Months Among YMSM at 12 Months
Description: as for outcome 6
Time Frame: Assessed at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mpowerment-based Intervention | Standard of Care
Number analyzed (Participants) | 234 | 231
Participants | 24 | 40

9. Primary Outcome: Prevalence of Condomless Anal Sex in the Past 6 Months Among YMSM at 18 Months
Description: as for outcome 6
Time Frame: Assessed at 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mpowerment-based Intervention | Standard of Care
Number analyzed (Participants) | 218 | 223
Participants | 29 | 39

10. Primary Outcome: Prevalence of Condomless Anal Sex in the Past 6 Months Among YMSM at 24 Months
Description: as for outcome 6
Time Frame: Assessed at 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mpowerment-based Intervention | Standard of Care
Number analyzed (Participants) | 187 | 205
Participants | 25 | 37

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a period of 24-months.
Arm/Group | Mpowerment-based Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/318 | 0/318
Serious Adverse Events (participants affected / at risk) | 0/318 | 0/318
Other Adverse Events (participants affected / at risk) | 0/318 | 0/318

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-01-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT05161689/Prot_SAP_ICF_000.pdf